CLINICAL TRIAL: NCT06215716
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Efruxifermin in Subjects With Non-Cirrhotic Nonalcoholic Steatohepatitis (NASH)/Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Fibrosis
Brief Title: A Study Evaluating Efruxifermin in Subjects With Non-Cirrhotic Nonalcoholic Steatohepatitis (NASH)/Metabolic Dysfunction-Associated Steatohepatitis (MASH) and Fibrosis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Akero Therapeutics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AK-US-001-0105
Record Dates: First submitted 2023-12-06; First posted 2024-01-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: NASH With Fibrosis; MASH With Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EFX 28 mg (Experimental)
  Interventions: Drug: Efruxifermin
- EFX 50 mg (Experimental)
  Interventions: Drug: Efruxifermin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efruxifermin — Administered by subcutaneous injection
  Arms: EFX 28 mg; EFX 50 mg
Drug: Placebo — Administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a multi-center evaluation of efruxifermin (EFX) in a randomized, double-blind, placebo-controlled study in subjects with non-cirrhotic NASH/MASH and fibrosis stage 2 or 3 (F2 or F3).

The study will enroll subjects in two cohorts for a total samples size of 1650 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant, non-lactating females between 18 - 80 years of age inclusive, based on the date of the screening visit.
* Previous history or presence of 2 out of 4 components of metabolic syndrome (obesity, dyslipidemia, elevated blood pressure, elevated fasting glucose) or type 2 diabetes.
* Cohort 1: Biopsy-proven NASH/MASH. Must have had a liver biopsy obtained ≤ 180 days prior to screening with fibrosis stage 2 or 3 and a non-alcoholic fatty liver disease (NAFLD) activity score (NAS) of ≥ 4 with at least a score of 1 in each of the following NAS components:

  * Steatosis (scored 0 to 3),
  * Ballooning degeneration (scored 0 to 2), and
  * Lobular inflammation (scored 0 to 3).

Exclusion Criteria:

* Other causes of liver disease based on medical history and/or liver histology and/or central laboratory results.
* Presence of cirrhosis on liver biopsy (fibrosis stage 4).
* Type 1 or uncontrolled Type 2 diabetes.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1650 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2032-11 (Estimated); Study Completion 2032-11 (Estimated)

PRIMARY OUTCOMES:
Cohort 1 Only: Resolution of NASH/MASH and a ≥ 1 stage improvement in fibrosis | 52 Weeks
  Based on NAS (scored by 0-1 for steatosis, 0-3 for inflammation, and 0-2 for ballooning) and NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)
Event-free survival | 240 Weeks
  Based on time from randomization to the first clinical event including evidence of disease progression, liver decompensation events, liver transplantation or eligibility for liver transplantation, and all-cause mortality.

SECONDARY OUTCOMES:
Cohort 1 Only: Resolution of NASH/MASH and no worsening of fibrosis | 52 Weeks
  Based on NAS (scored by 0-1 for steatosis, 0-3 for inflammation, and 0-2 for ballooning) and NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)
Cohort 1 Only: ≥ 1 stage improvement in fibrosis and no worsening of steatohepatitis | 52 Weeks
  Based on NAS (scored by 0-1 for steatosis, 0-3 for inflammation, and 0-2 for ballooning) and NASH CRN fibrosis score (scored by a fibrosis score of 0-4, where 0 = no fibrosis, 1 = centrilobular pericellular fibrosis, 2 = centrilobular and periportal fibrosis, 3 = bridging fibrosis, 4 = cirrhosis)
Change from baseline of non-invasive markers of liver fibrosis | 52 Weeks, 240 Weeks
  ELF (scale of 6.7 to 9.8 when higher scores indicative of increased fibrosis)
Change from baseline of non-invasive markers of liver fibrosis | 52 Weeks, 240 Weeks
  Pro-C3 (ug/L)
Change from baseline of non-invasive markers of liver fibrosis | 52 Weeks, 240 Weeks
  Liver stiffness assessed by transient elastography (FibroScan®) (kPa, CAP)
Change from baseline of markers of liver injury | 52 Weeks, 240 Weeks
  ALT (U/L), AST (U/L), GGT (U/L)
Change from baseline of markers of liver injury | 52 Weeks, 240 Weeks
  Uric acid (mg/dL)
Change from baseline of lipoproteins | 52 Weeks, 240 Weeks
  Total cholesterol (mg/dL), TG (mg/dL), Non-HDL-C (mg/dL), HDL-C (mg/dL), and LDL-C (mg/dL)
Change from baseline of markers of insulin sensitivity and glycemic control | 52 Weeks, 240 Weeks
  HbA1c (%)
Change from baseline of markers of insulin sensitivity and glycemic control | 52 Weeks, 240 Weeks
  Adiponectin (mg/L)
Change from baseline of body weight (kg) | 52 Weeks, 240 Weeks
To assess the safety and tolerability of EFX through the reporting of extent of exposure (weeks) | 52 Weeks, 240 Weeks
To assess the safety and tolerability of EFX through the reporting of adverse events (severity of events) | 52 Weeks, 240 Weeks
To assess the safety and tolerability of EFX through the reporting of adverse events (frequency of events) | 52 Weeks, 240 Weeks
To assess the safety and tolerability of EFX through the reporting of abnormal clinical laboratory tests, ECGs, ultrasounds, vital sign assessments (number of patients) | 52 Weeks, 240 Weeks
To assess the immunogenicity of EFX through the reporting of antidrug antibodies (number of patients) | 52 Weeks, 240 Weeks

CONTACTS AND LOCATIONS:
Locations (278):
- United States (160):
  - Akero Clinical Study Site, Birmingham, Alabama
  - Akero Clinical Study Site, Dothan, Alabama
  - Akero Clinical Study Site, Chandler, Arizona
  - Akero Clinical Study Site, Flagstaff, Arizona
  - Akero Clinical Study Site, Mesa, Arizona
  - Akero Clinical Study Site, Peoria, Arizona
  - Akero Clinical Study Site, Tucson, Arizona
  - Akero Clinical Study Site, Conway, Arkansas
  - Akero Clinical Study Site, Jonesboro, Arkansas
  - Akero Clinical Study Site, Little Rock, Arkansas
  - Akero Clinical Study Site, North Little Rock, Arkansas
  - Akero Clinical Study Site, Chula Vista, California
  - Akero Clinical Study Site, Coronado, California
  - Akero Clinical Study Site, Escondido, California
  - Akero Clinical Study Site, Folsom, California
  - Akero Clinical Study Site, Inglewood, California
  - Akero Clinical Study Site, La Mesa, California
  - Akero Clinical Study Site, Lancaster, California
  - Akero Clinical Study Site, Long Beach, California
  - Akero Clinical Study Site, Los Angeles, California
  - Akero Clinical Study Site, Newport Beach, California
  - Akero Clinical Study Site, Orange, California
  - Akero Clinical Study Site, Palm Springs, California
  - Akero Clinical Study Site, Pasadena, California
  - Akero Clinical Study Site, Redwood City, California
  - Akero Clinical Study Site, San Diego, California
  - Akero Clinical Study Site, San Francisco, California
  - Akero Clinical Study Site, Santa Maria, California
  - Akero Clinical Study Site, Aurora, Colorado
  - Akero Clinical Study Site, Colorado Springs, Colorado
  - Akero Clinical Study Site, Englewood, Colorado
  - Akero Clinical Study Site, New Haven, Connecticut
  - Akero Clinical Study Site, Washington D.C., District of Columbia
  - Akero Clinical Study Site, Bradenton, Florida
  - Akero Clinical Study Site, Brandon, Florida
  - Akero Clinical Study Site, Doral, Florida
  - Akero Clinical Study Site, Fort Myers, Florida
  - Akero Clinical Study Site, Gainesville, Florida
  - Akero Clinical Study Site, Hialeah Gardens, Florida
  - Akero Clinical Study Site, Inverness, Florida
  - Akero Clinical Study Site, Jacksonville, Florida
  - Akero Clinical Study Site, Lady Lake, Florida
  - Akero Clinical Study Site, Lakewood Rch, Florida
  - Akero Clinical Study Site, Largo, Florida
  - Akero Clinical Study Site, Lehigh Acres, Florida
  - Akero Clinical Study Site, Maitland, Florida
  - Akero Clinical Study Site, Margate, Florida
  - Akero Clinical Study Site, Miami, Florida
  - Akero Clinical Study Site, Miami Gardens, Florida
  - Akero Clinical Study Site, Miami Lakes, Florida
  - Akero Clinical Study Site, Naples, Florida
  - Akero Clinical Study Site, New Port Richey, Florida
  - Akero Clinical Study Site, Ocala, Florida
  - Akero Clinical Study Site, Orlando, Florida
  - Akero Clinical Study Site, Pembroke Pines, Florida
  - Akero Clinical Study Site, Port Orange, Florida
  - Akero Clinical Study Site, Riverview, Florida
  - Akero Clinical Study Site, Sarasota, Florida
  - Akero Clinical Study Site, Temple Terrace, Florida
  - Akero Clinical Study Site, Venice, Florida
  - Akero Clinical Study Site, Viera, Florida
  - Akero Clinical Study Site, West Palm Beach, Florida
  - Akero Clinical Study Site, Winter Park, Florida
  - Akero Clinical Study Site, Zephyrhills, Florida
  - Akero Clinical Study Site, Atlanta, Georgia
  - Akero Clinical Study Site, Columbus, Georgia
  - Akero Clinical Study Site, Gainesville, Georgia
  - Akero Clinical Study Site, Marietta, Georgia
  - Akero Clinical Study Site, Chicago, Illinois
  - Akero Clinical Study Site, Hammond, Indiana
  - Akero Clinical Study Site, Indianapolis, Indiana
  - Akero Clinical Study Site, South Bend, Indiana
  - Akero Clinical Study Site, West Des Moines, Iowa
  - Akero Clinical Study Site, Topeka, Kansas
  - Akero Clinical Study Site, Wichita, Kansas
  - Akero Clinical Study Site, Louisville, Kentucky
  - Akero Clinical Study Site, Bastrop, Louisiana
  - Akero Clinical Study Site, Covington, Louisiana
  - Akero Clinical Study Site, Houma, Louisiana
  - Akero Clinical Study Site, Marrero, Louisiana
  - Akero Clinical Study Site, Metairie, Louisiana
  - Akero Clinical Study Site, New Orleans, Louisiana
  - Akero Clinical Study Site, Shreveport, Louisiana
  - Akero Clinical Study Site, West Monroe, Louisiana
  - Akero Clinical Study Site, Baltimore, Maryland
  - Akero Clinical Study Site, Glen Burnie, Maryland
  - Akero Clinical Study Site, Greenbelt, Maryland
  - Akero Clinical Study Site, South Dartmouth, Massachusetts
  - Akero Clinical Study Site, Novi, Michigan
  - Akero Clinical Study Site, Southfield, Michigan
  - Akero Clinical Study Site, Wyoming, Michigan
  - Akero Clinical Study Site, Ypsilanti, Michigan
  - Akero Clinical Study Site, Flowood, Mississippi
  - Akero Clinical Study Site, Columbia, Missouri
  - Akero Clinical Study Site, Kansas City, Missouri
  - Akero Clinical Study Site, St Louis, Missouri
  - Akero Clinical Study Site, Las Vegas, Nevada
  - Akero Clinical Study Site, Reno, Nevada
  - Akero Clinical Study Site, Florham Park, New Jersey
  - Akero Clinical Study Site, Ridgewood, New Jersey
  - Akero Clinical Study Site, Somers Point, New Jersey
  - Akero Clinical Study Site, Sparta, New Jersey
  - Akero Clinical Study Site, Santa Fe, New Mexico
  - Akero Clinical Study Site, Buffalo, New York
  - Akero Clinical Study Site, New York, New York
  - Akero Clinical Study Site, Rochester, New York
  - Akero Clinical Study Site, Chapel Hill, North Carolina
  - Akero Clinical Study Site, Charlotte, North Carolina
  - Akero Clinical Study Site, Durham, North Carolina
  - Akero Clinical Study Site, Fayetteville, North Carolina
  - Akero Clinical Study Site, Morehead City, North Carolina
  - Akero Clinical Study Site, New Bern, North Carolina
  - Akero Clinical Study Site, Raleigh, North Carolina
  - Akero Clinical Study Site, Statesville, North Carolina
  - Akero Clinical Study Site, Columbus, Ohio
  - Akero Clinical Study Site, Dayton, Ohio
  - Akero Clinical Study Site, Springboro, Ohio
  - Akero Clinical Study Site, Westlake, Ohio
  - Akero Clinical Study Site, Medford, Oregon
  - Akero Clinical Study Site, Hershey, Pennsylvania
  - Akero Clinical Study Site, Philadelphia, Pennsylvania
  - Akero Clinical Study Site, Pittsburgh, Pennsylvania
  - Akero Clinical Study Site, Charleston, South Carolina
  - Akero Clinical Study Site, Columbia, South Carolina
  - Akero Clinical Study Site, Summerville, South Carolina
  - Akero Clinical Study Site, Chattanooga, Tennessee
  - Akero Clinical Study Site, Clarksville, Tennessee
  - Akero Clinical Study Site, Hermitage, Tennessee
  - Akero Clinical Study Site, Nashville, Tennessee
  - Akero Clinical Study Site, Amarillo, Texas
  - Akero Clinical Study Site, Austin, Texas
  - Akero Clinical Study Site, Bellaire, Texas
  - Akero Clinical Study Site, Brownsville, Texas
  - Akero Clinical Study Site, Corpus Christi, Texas
  - Akero Clinical Study Site, Dallas, Texas
  - Akero Clinical Study Site, Denison, Texas
  - Akero Clinical Study Site, Edinburg, Texas
  - Akero Clinical Study Site, Forney, Texas
  - Akero Clinical Study Site, Fort Worth, Texas
  - Akero Clinical Study Site, Houston, Texas
  - Akero Clinical Study Site, Lewisville, Texas
  - Akero Clinical Study Site, McAllen, Texas
  - Akero Clinical Study Site, Pasadena, Texas
  - Akero Clinical Study Site, San Antonio, Texas
  - Akero Clinical Study Site, San Marcos, Texas
  - Akero Clinical Study Site, Waco, Texas
  - Akero Clinical Study Site, Webster, Texas
  - Akero Clinical Study Site, Wichita Falls, Texas
  - Akero Clinical Study Site, Ogden, Utah
  - Akero Clinical Study Site, Salt Lake City, Utah
  - Akero Clinical Study Site, Sandy City, Utah
  - Akero Clinical Study Site, South Ogden, Utah
  - Akero Clinical Study Site, Falls Church, Virginia
  - Akero Clinical Study Site, Newport News, Virginia
  - Akero Clinical Study Site, Norfolk, Virginia
  - Akero Clinical Study Site, Richmond, Virginia
  - Akero Clinical Study Site, Roanoke, Virginia
  - Akero Clinical Study Site, Suffolk, Virginia
  - Akero Clinical Study Site, Seattle, Washington
  - Akero Clinical Study Site, Spokane, Washington
- Argentina (5):
  - Akero Clinical Study Site, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Akero Clinical Study Site, La Plata, Buenos Aires
  - Akero Clinical Study Site, Ramos Mejía, Buenos Aires
  - Akero Clinical Study Site, Buenos Aires, Distrito Federal
  - Akero Clinical Study Site, Buenos Aires
- Australia (13):
  - Akero Clinical Study Site, Broadmeadow, New South Wales
  - Akero Clinical Study Site, Kogarah, New South Wales
  - Akero Clinical Study Site, Liverpool, New South Wales
  - Akero Clinical Study Site, Westmead, New South Wales
  - Akero Clinical Study Site, Adelaide, South Australia
  - Akero Clinical Study Site, Caulfield South, Victoria
  - Akero Clinical Study Site, Epping, Victoria
  - Akero Clinical Study Site, Frankston, Victoria
  - Akero Clinical Study Site, Heidelberg, Victoria
  - Akero Clinical Study Site, Melbourne, Victoria
  - Akero Clinical Study Site, Murdoch, Western Australia
  - Akero Clinical Study Site, Nedlands, Western Australia
  - Akero Clinical Study Site, Perth, Western Australia
- Canada (6):
  - Akero Clinical Study Site, Edmonton, Alberta
  - Akero Clinical Study Site, Hamilton, Ontario
  - Akero Clinical Study Site, Toronto, Ontario
  - Akero Clinical Study Site, Vaughan, Ontario
  - Akero Clinical Study Site, Montreal, Quebec
  - Akero Clinical Study Site, Terrebonne, Quebec
- France (12):
  - Akero Clinical Study Site, Nice, Alpes-Maritimes
  - Akero Clinical Study Site, Lyon, Auvergne-Rhône-Alpes
  - Akero Clinical Study Site, Strasbourg, Bas-Rhin
  - Akero Clinical Study Site, Limoges, Haute-Vienne
  - Akero Clinical Study Site, Clichy, Hauts-de-Seine
  - Akero Clinical Study Site, Vandœuvre-lès-Nancy, Lorraine
  - Akero Clinical Study Site, Angers, Maine-et-Loire
  - Akero Clinical Study Site, Toulouse, Occitanie
  - Akero Clinical Study Site, Marseille, Provence-Alpes-Côte d'Azur Region
  - Akero Clinical Study Site, Montpellier Cedex 5, Provence-Alpes-Côte d'Azur Region
  - Akero Clinical Study Site, Versailles, Yvelines, Île-de-France
  - Akero Clinical Study Site, Paris, Île-de-France Region
- Germany (6):
  - Akero Clinical Study Site, Würzburg, Bavaria
  - Akero Clinical Study Site, Frankfurt am Main, Hesse
  - Akero Clinical Study Site, Mainz, Rhineland-Palatinate
  - Akero Clinical Study Site, Leipzig, Saxony
  - Akero Clinical Study Site, Lübeck, Schleswig-Holstein
  - Akero Clinical Study Site, Berlin
- India (12):
  - Akero Clinical Study Site, Surat, Gujarat
  - Akero Clinical Study Site, Vadodara, Gujarat
  - Akero Clinical Study Site, Thiruvananthapuram, Kerala
  - Akero Clinical Study Site, Dahegaon, Maharashtra
  - Akero Clinical Study Site, Nagpur, Maharashtra
  - Akero Clinical Study Site, Pune, Maharashtra
  - Akero Clinical Study Site, New Delhi, National Capital Territory of Delhi
  - Akero Clinical Study Site, Jaipur, Rajasthan
  - Akero Clinical Study Site, Coimbatore, Tamil Nadu
  - Akero Clinical Study Site, Hyderabad, Telangana
  - Akero Clinical Study Site, Varanasi, Uttar Pradesh
  - Akero Clinical Study Site, Kolkata, West Bengal
- Israel (8):
  - Akero Clinical Study Site, Petah Tikva, Central District
  - Akero Clinical Study Site, Ramat Gan, Central District
  - Akero Clinical Study Site, Haifa, Haifa District
  - Akero Clinical Study Site, Afula, Northern District
  - Akero Clinical Study Site, Nahariya, Northern District
  - Akero Clinical Study Site, Nazareth, Northern District
  - Akero Clinical Study Site, Jerusalem
  - Akero Clinical Study Site, Tel Aviv
- Italy (10):
  - Akero Clinical Study Site, San Giovanni Rotondo, Foggia
  - Akero Clinical Study Site, Rozzano, Milan
  - Akero Clinical Study Site, Torino, Turin
  - Akero Clinical Study Site, Bologna
  - Akero Clinical Study Site, Foggia
  - Akero Clinical Study Site, Messina
  - Akero Clinical Study Site, Milan
  - Akero Clinical Study Site, Modena
  - Akero Clinical Study Site, Napoli
  - Akero Clinical Study Site, Novara
- Akero Clinical Study Site, Cuauhtémoc, Mexico City, Mexico
- Poland (9):
  - Akero Clinical Study Site, Poznan, Greater Poland Voivodeship
  - Akero Clinical Study Site, Krakow, Lesser Poland Voivodeship
  - Akero Clinical Study Site, Wroclaw, Lower Silesian Voivodeship
  - Akero Clinical Study Site, Warsaw, Masovian Voivodeship
  - Akero Clinical Study Site, Gdansk, Pomeranian Voivodeship
  - Akero Clinical Study Site, Gdynia, Pomeranian Voivodeship
  - Akero Clinical Study Site, Częstochowa, Silesian Voivodeship
  - Akero Clinical Study Site, Katowice, Silesian Voivodeship
  - Akero Clinical Study Site, Lodz, Łódź Voivodeship
- Puerto Rico (3):
  - Akero Clinical Study Site, Manatí
  - Akero Clinical Study Site, Mayagüez
  - Akero Clinical Study Site, San Juan
- South Korea (7):
  - Akero Clinical Study Site, Daegu, Daegu Gwang'yeogsi [Taegu-Kwangyokshi]
  - Akero Clinical Study Site, Goyang-si, Gyeonggi-do
  - Akero Clinical Study Site, Incheon, Gyeonggi-do
  - Akero Clinical Study Site, Seongnam-si, Gyeonggi-do
  - Akero Clinical Study Site, Seongnam-si, Gyeonggido [Kyonggi-do]
  - Akero Clinical Study Site, Daegu, Gyeongsangbugdo [Kyongsangbuk-do]
  - Akero Clinical Study Site, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
- Spain (7):
  - Akero Clinical Study Site, Sabadell, Barcelona
  - Akero Clinical Study Site, Santander, Cantabria
  - Akero Clinical Study Site, Majadahonda, Madrid
  - Akero Clinical Study Site, Valencia, València
  - Akero Clinical Study Site, Barcelona
  - Akero Clinical Study Site, Madrid
  - Akero Clinical Study Site, Seville
- Switzerland (3):
  - Akero Clinical Study Site, Olten, Canton of Solothurn
  - Akero Clinical Study Site, Bern
  - Akero Clinical Study Site, Sankt Gallen
- Taiwan (7):
  - Akero Clinical Study Site, Changhua, Changhua
  - Akero Clinical Study Site, Taichung, Taichung
  - Akero Clinical Study Site, Tainan, Tainan
  - Akero Clinical Study Site, Taipei City, Taipei
  - Akero Clinical Study Site, Kaohsiung City
  - Akero Clinical Study Site, Tainan
  - Akero Clinical Study Site, Taoyuan District
- Turkey (Türkiye) (4):
  - Akero Clinical Study Site, Yenimahalle, Ankara
  - Akero Clinical Study Site, Bornova, İzmir
  - Akero Clinical Study Site, Bursa
  - Akero Clinical Study Site, Rize
- United Kingdom (5):
  - Akero Clinical Study Site, Birmingham, England
  - Akero Clinical Study Site, Cambridge, England
  - Akero Clinical Study Site, Liverpool, England
  - Akero Clinical Study Site, London, England
  - Akero Clinical Study Site, Newcastle upon Tyne, England

IPD SHARING:
Plan to Share IPD: No